CLINICAL TRIAL: NCT01630954
Title: A Comparison of Single Versus Double Evacuation for Treatment of Hydatidiform
Brief Title: A Comparison of Single Versus Double Evacuation for Treatment of Hydatidiform Mole
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nilratan Sircar Medical College (Other Government)
Responsible Party: Principal Investigator, Dr Snehamay Chaudhuri, Associate Professor,Obstetrics and Gynecology, NRS Medical College, Nilratan Sircar Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-Chaudhuri
Record Dates: First submitted 2012-06-24; First posted 2012-06-28 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Hydatidiform Mole
Keywords: Hydatidiform mole; Molar pregnancy; H Mole; GTN; GTD
MeSH Terms: conditions — Hydatidiform Mole | interventions — Suction; Vacuum Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single evacuation of mole, (Active Comparator)
  Interventions: Procedure: Suction and evacuation
- Double evacuation of mole (Active Comparator)
  Interventions: Procedure: Suction and evacuation

INTERVENTIONS:
Procedure: Suction and evacuation — In single evacuation group women will be treated by suction evacuation and curettage is performed at the end of evacuation in one sitting. An ultrasound will be done later to examine completeness of evacuation. If there is significant amount of residual molar tissue or persistence of heavy bleeding a repeat curettage will be done . Women will be followed up with serum beta hcg 1 week after the evacuation and then weekly till the titer is negative. After three consecutive negative titre beat HCG estimation will be done at two weekly interval.
  Other Names: Suction curettage
  Arms: Single evacuation of mole,
Procedure: Suction and evacuation — In double evacuation group , women will be treated by suction evacuation and a thorough curettage will be avoided. A second evacuation with thorough curettage will be performed after 5 - 7 days of first evacuation.
  Other Names: Suction curettage
  Arms: Double evacuation of mole

SUMMARY:
Hydatidiform mole is a common complication of pregnancy with an incidence of 1in 400 pregnancies in India. Although this is a benign condition , it is having the malignant potential too. A repeat curettage after evacuation of hydatidiform mole was generally advocated till 1990s. A thorough curettage at the time of initial evacuation was not performed because of larger size of uterus and risk of perforation. Subsequently a number of studies assessed the usefulness of repeat curettage and found it was unnecessary and not cost effective . However all these studies are retrospective in design and conducted in developed countries where hydatidiform mole is diagnosed earlier because of wider use of ultrasonography. Thus there is a need to perform a well designed prospective study to compare the effectiveness of single evacuation with double evacuation in treatment of hydatidiform mole for prevention of Gestational Trophoblastic Neoplasia.This study compares the effectiveness of single evacuation versus double evacuation for treatment of hydatidiform mole for prevention of gestational trophoblastic neoplasia .

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound confirmed complete mole

Exclusion Criteria:

* Partial mole
* History of treatment for molar pregnancy like prior evacuation or chemotherapy
* Women requiring hysterectomy for treatment of H Mole

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patents diagnosed as GTN following treatment in each group | Six months following evacuation

SECONDARY OUTCOMES:
Maternal complications, | Six months
Time interval of normalization of HCG | Six months following evacuation
Duration of hospital stay | Two weeks following admission

CONTACTS AND LOCATIONS:
Overall Officials: Snehamay Chaudhuri, MD, DNB, Principal Investigator — Associate Professor, Obstetrics and Gynecology, NRS Medical College , Kolkata,India
Locations (1):
- Dr Snehamay Chaudhuri, Kolkata, West Bengal, India